CLINICAL TRIAL: NCT05734950
Title: Biological Characteristics of Older Women (> 70 Years) With Oestrogen-receptor (ER) Positive, Human Epidermal Growth Factor 2 (HER2) Negative Early Breast Cancer: Definition of Molecular and Genomic Features.
Brief Title: Biological Characteristics of Older Women (> 70 Years) With ER Positive, HER2 Negative Early Breast Cancer
Acronym: BOLD-70
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Institute of Cancer Research, United Kingdom (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: CCR5654
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Translational study — Non-interventional, translational study

SUMMARY:
This study is investigating the biological characteristics of early oestrogen receptor (ER) positive, human epidermal growth factor receptor 2 (HER2) negative breast cancer (BC) in older woman (aged > 70 years) who were treated with adjuvant endocrine treatment (ET). It will use surgical tissue previously collected as part of routine care from patients aged 70 years or older at diagnosis with ER positive, HER2 negative stage I-III BC treated The Royal Marsden NHS Foundation Trust (RMH).

The overarching aim of this study is to define the biological characteristics of early BC in older women in terms of tumour microenvironment (TME), molecular and genomic features. This analysis will include assessment of tumour infiltrating lymphocytes (TILs), and gene expression profiling with NanoString using the Breast Cancer 360 (BC360TM) assay measuring ribonucleic acid (RNA) expression signatures of genes involved in proliferation, endothelial, angiogenesis, cytotoxicity, stroma, inflammatory chemokines, and apoptosis. This analysis will examine various biological pathways, aiming to inform suitability for certain treatments including cyclin-dependent kinase inhibitors (CDKi), chemotherapy, immunotherapy, or targeted treatments such as phosphoinositide 3-kinases (PI3K) inhibitors, or deoxyribonucleic acid (DNA) damage response.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women aged >70 years at the time of diagnosis of invasive breast cancer.
* ER positive (Allred score >5/8), HER2 negative early invasive BC.
* Stage I-III BC.
* Surgical tissue available.
* No pre-surgical systemic therapy (i.e., no pre-operative ET or chemotherapy).
* Planned adjuvant ET with an aromatase-inhibitor.
* No adjuvant chemotherapy.
* Surgery was performed between 1st January 2014 and 31st December 2016.

Exclusion Criteria:

* Pre- or perimenopausal.
* ER negative or HER2-positive BC.
* Multifocal cancer where not all of foci ER positive HER2 negative
* Bilateral breast cancer.
* Stage IV breast cancer.
* Benign histology or DCIS.
* Pre-surgical treatment.
* Prior chemotherapy for BC.

Min Age: 71 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes
Study Population: This is a non-interventional, translational study, using surgical tissue (collected as part of routine care) from older women (aged > 70 years at the time of diagnosis) with early (stage I-III), ER positive, HER2 negative BC who were treated curatively with primary surgery. Patients would not have had any prior treatment with (neo-) adjuvant chemotherapy but received an aromatase-inhibitor in the adjuvant setting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Distribution of TILs percentage | August 2023
  assessed via immunohistochemistry

SECONDARY OUTCOMES:
Gene expression profile patterns across the cohort. | August 2023
  assessed via genomic profiling
Relationship between PAM50, Ki67 (<10% low, ≥ 10% high), PD-L1, modified AIR-CIS | August 2023
  assessed with advanced machine learning methods

OTHER OUTCOMES:
Association of the molecular features with TTR (Defined as the time from diagnosis (initial biopsy) to local, regional, or distant tumour recurrence or death from breast cancer without prior notification of relapse.). | August 2023
  Exploratory

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No